CLINICAL TRIAL: NCT00613808
Title: An Investigation of Topical Application of Gaseous Nitric Oxide on Safety and Efficacy in Venous Stasis Ulcers of the Lower Extremities
Brief Title: Safety and Efficacy of Gaseous Nitric Oxide on Venous Stasis Leg Ulcers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Nitric BioTherapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP 3
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Venous Ulcers
Keywords: venous; leg; ulcer
MeSH Terms: conditions — Varicose Ulcer; Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A - Standard of Care (control) (No Intervention): Standard of care - dressings and sustained compression only for the two week screening period and then for 20 weeks thereafter
- B Same treatment for 6 weeks, 200ppm NO gas (Active Comparator): Subjects were treated by topical application of 200ppm Nitric Oxide gas delivered to the wound area for 8 hours per day for 6 weeks
  Interventions: Drug: Nitric Oxide 200ppm Group B

INTERVENTIONS:
Drug: Nitric Oxide 200ppm Group B — 200 ppm, 8hrs / day for 6 weeks
  Arms: B Same treatment for 6 weeks, 200ppm NO gas

SUMMARY:
The purpose of this study is to determine whether nitric oxide (NO)gas is effective in the treatment of venous ulcers of the lower leg.

DETAILED DESCRIPTION:
SUbjects were divided into two Groups - one receiving 200ppm NO gas delivered topically to the wound area for 8 hours a day for 6 weeks. The other Group (control arm) received Standard of Care (compression) for 22 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must have given written informed consent and HIPAA authorization
* Must be ≥ 18 years of age
* Must have a venous ulcer for 60 days or greater
* ABPI > 0.8 and ≤ 1.2
* Must have ulcer between 3cm2 and 25cm2 in size

Exclusion Criteria:

* Has an ulcer that is deemed by the Investigator to be caused primarily by a medical condition other than venous insufficiency
* BMI ≥ 35
* Has evidence of clinical infection
* Suffers from diabetes mellitus with HbA1c ≥ 8%
* Suffers from clinically significant arterial disease
* Has a known allergy to any of the compounds / drugs that are part of this protocol
* Has evidence of the ulcer and / or infection extending to the underlying muscle, tendon or bone
* Has used any investigational drug(s) within 30 days preceding randomization
* Is unable to manage self-treatment
* Is pregnant, nursing mother or a woman of child bearing potential who is not using an adequate form of contraception (or abstinence)
* Suffers from a condition which in the opinion of the Investigator would compromise the safety of the subject and / or the quality of the data
* Is using any of the prohibited concomitant medications or treatments
* Has previously participated in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Effect of daily application of Nitric Oxide on rate of closure in venous ulcers | 24 weeks or wound closure

SECONDARY OUTCOMES:
Change in quality of life | 24 weeks or wound closure
Incidence of adverse events | 24 weeks or wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Jensen, DPM, Principal Investigator — Private Practice, Denver, CO
Locations (2):
- United States (2):
  - Diabetic Foot & Wound Center, Denver, Colorado
  - Alamo Podiatry Associates, San Antonio, Texas